CLINICAL TRIAL: NCT04568577
Title: Effects of the Elastic Taping on the Chronic Ankle Instability: a Clinical Trial
Brief Title: Effects of the Elastic Taping on the Chronic Ankle Instability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Norte do Paraná (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 3.059.113
Record Dates: First submitted 2020-05-14; First posted 2020-09-29 (Actual); Last update posted 2020-09-29 (Actual); Status verified 2020-09

CONDITIONS: Ankle Sprains; Chronic Ankle Instability; Athletes Foot
Keywords: Athletic Tape; Ankle Sprains; Chronic Ankle Instability
MeSH Terms: conditions — Ankle Injuries; Tinea Pedis | interventions — Compression Bandages

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- tensioned tape (Experimental): The tensioned tape group will apply weekly with gradual tension calculated by measuring the initial length of the tape. From the first week of application, there will be a 5% increase in tension up to the fifth week.
  Interventions: Other: Tape with tension
- tape without tension (Active Comparator): The tensionless tape group will receive the application of the tape weekly without tensioning during the five weeks.
  Interventions: Other: Tape without tension

INTERVENTIONS:
Other: Tape with tension — The elastic bandage will be applied with a voltage increase controlled weekly, for five weeks. Each week, 5% of tension will be added to the application. In the first week the application will be tension-free.
  Other Names: Elastic tape; Kinesiotaping; Tape tensioned; Elastic bandage
  Arms: tensioned tape
Other: Tape without tension — Bandaging applications will be weekly, for five weeks, without tensioning the tape.
  Other Names: elastic tape; elastic bandage; kinesiotaping
  Arms: tape without tension

SUMMARY:
This study will analyze the effects of an elastic taping application protocol in individuals with chronic ankle instability. One group will perform a protocol with increased tape tension for five weeks while the other group will receive the same tape without tension during the same period.

DETAILED DESCRIPTION:
Elastic taping is a method widely used in clinical practice for the treatment of ankle instability and shows increasing interest in research to verify its effectiveness. The literature presents several studies with short-term effects, largely in healthy individuals and with several application techniques, with the incremental tensioning of the proposed tape subjectively.

The literature presents several studies with short-term effects, largely in healthy individuals and with several application techniques, with the incremental tensioning of the proposed tape subjectively.

ELIGIBILITY:
Inclusion Criteria:

* young adults with chronic ankle instability (unilateral or bilateral);
* the first sprain episode occurred for at least 1 year pre-study associated with inflammatory symptoms (pain, edema, etc.);
* having discontinued for at least 1 day physical activity;
* the most recent sprain occurred more than 3 months prior study;
* self-reported instability feeling to be confirmed by specific questionnaires.

Exclusion Criteria:

* lower limb surgical procedure;
* lower limb fracture history;
* acute injury (last 3 months) of other lower limb joints resulting in at least 1 day in the interruption of physical activity;
* wounds in the ankle region or foot;
* own skin disease;
* have allergy to bandage;
* be in physiotherapeutic treatment.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2019-06-24 (Actual); Study Completion 2019-08-26 (Actual)

PRIMARY OUTCOMES:
Functionality | The evaluation will occur at week 1 (baseline) and at the end of the protocol (week 6)
  The functionality will be evaluated by the average of three executions of the side hop test and dynamic balance test (star excursion balance test modified). The side hop test consists of lateral jumps beyond the 30 cm mark on the ground in the shortest possible time (the shorter the time, the better the performance). The dynamic balance test consists of remaining in unipodal support and reaching as far as possible with the other member in the anterior, posteromedial and posterolateral directions. The greater the distance achieved improves the score. The calculation is performed to correct the measurements.

SECONDARY OUTCOMES:
Balance | The evaluation will occur at week 1 (baseline) and at the end of the protocol (week 6)
  The balance will be evaluated by the force platform at baseline. The variables center of pressure, speed of displacement of the center of pressure in the anteroposterior and mediolateral directions, frequency of displacement of the center of pressure in the anteroposterior and mediolateral directions will be analyzed. The lower the score, the better the performance.
Self-reported instability | The evaluation will occur at week 1 (baseline) and at the end of the protocol (week 6)
  Self-reported instability will be assessed by questionnaire. The Cumberland Ankle Instability Tool consists of 9 questions with a maximum score of 30 points. Ankle instability is considered to have a score less than or equal to 24. The lower the score, the worse the instability. The other questionnaire used will be Foot and Ankle Outcome Score, which has 42 questions divided into 5 domains. Each domain has a score of 100%. If the individual has <75% in 3 domains, he is considered to have functional ankle instability. The lower the score, the worse the instability.

CONTACTS AND LOCATIONS:
Overall Officials: Gustavo FM Oliveira, researcher, Principal Investigator — Universidade Norte do Paraná
Locations (1):
- Gustavo Felipe Marques de Oliveira, Londrina, Paraná, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Miklovic TM, Donovan L, Protzuk OA, Kang MS, Feger MA. Acute lateral ankle sprain to chronic ankle instability: a pathway of dysfunction. Phys Sportsmed. 2018 Feb;46(1):116-122. doi: 10.1080/00913847.2018.1409604. Epub 2017 Nov 29. PMID 29171312
- [Result] Delahunt E, Remus A. Risk Factors for Lateral Ankle Sprains and Chronic Ankle Instability. J Athl Train. 2019 Jun;54(6):611-616. doi: 10.4085/1062-6050-44-18. Epub 2019 Jun 4. PMID 31161942

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-22): https://cdn.clinicaltrials.gov/large-docs/77/NCT04568577/Prot_SAP_000.pdf